CLINICAL TRIAL: NCT06860906
Title: Outcome of V-Y Anoplasty Techniques in Management of Anal Stenosis
Brief Title: V-Y Flap for Anal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #11393-17-12-2023
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-12

CONDITIONS: Anal Stenosis
Keywords: anal stenosis, anoplasty, V-Y advancement flap
MeSH Terms: conditions — Anus, Imperforate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with anal stenosis (Experimental)
  Interventions: Procedure: V-Y advancement flap

INTERVENTIONS:
Procedure: V-Y advancement flap — anal stenosis treated by removal of scarring tissue and cover the defect using V-Y advancement flap

SUMMARY:
anal stenosis is a common complication after massive open hemorrhoidectomy. it interferes with the patient daily activities. Many interventions were described, but there is no standard treatment. Data were always lost about the best intervention. In this study we try to discover if V-Y advancement flap can effectively treat anal stenosis or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 18years old with moderate to severe post- hemorrhoidectomy anal stenosis

Exclusion Criteria:

* pregnant females
* patient with prior radiation
* patient with T.B
* Patient with Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
operative time | Intraoperative (operative time is measured in minutes from incision to wound dressing)
pain score | from one day to 6 months postoperative
  pain score was measured by visual analogue scale. maximum value 10 indicated very painful while minimum value 0 meant painless
bleeding amount | from incision to 2 weeks after surgery
  intra and post operative bleeding amount is measured in cc by volumetric method
post-operative analgesia | from one day to 2 weeks post operative
  analgesia doses requirements of NSAIDs were measured in ml
hospital stay | for 1 to 2 days after surgery
  the duration of hospital stay was measured in days
healing time | healing duration in days calculated from the first day post operative to 3 months
  healing time was measured in days

SECONDARY OUTCOMES:
age | for 2 days before surgery
  age was recorded in years
sex | 2 days pre-operative
  sex (male or female) was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
data will be available on demand by contacting the principle investigator